CLINICAL TRIAL: NCT02614521
Title: A Single-center, Observational, 12-months Study to Examine the Predictive Factors for Successful Outcome After Pulmonary Veins Ablation to Treat Patients With Paroxysmal Atrial Fibrillation.
Brief Title: Predictive Factors for Successful Outcome After Pulmonary Veins Ablation to Treat Paroxysmal Atrial Fibrillation
Status: Withdrawn | Type: Observational
Sponsor: Elpen Pharmaceutical Co. Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 2015-IIS-GR-AF
Record Dates: First submitted 2015-11-23; First posted 2015-11-25 (Estimated); Last update posted 2019-05-13 (Actual); Status verified 2018-12

CONDITIONS: Atrial Fibrillation
Keywords: Pulmonary veins ablation; Paroxysmal atrial fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: pulmonary veins ablation's successful outcome — Assessment of predictive factors in patients with successful outcome of pulmonary veins ablations and suffer from paroxysmal atrial fibrillation.

SUMMARY:
Atrial fibrillation is the most common serious abnormal heart rhythm affecting about 2% to 3% of the population, being associated with a 1.5- to 1.9-fold higher risk of death. Patients with paroxysmal AF in whom antiarrhythmic drug therapy does not elicit a response are potential candidates for RF ablation of AF. The success rate of RF ablation in the treatment of AF varies depending on the type and duration of AF (ie, paroxysmal vs persistent), structural remodeling of the heart, co-morbidities and the technique of the cardiac electrophysiologist, but it usually ranges from 60-80% over 1-2 years of follow-up.

To study and predict the successful outcome of RF ablation is of great clinical importance. Moreover, the detection of predictive factors for successful outcome may alter the therapeutic strategy determining a subgroup of patients in the need of more invasive management.

DETAILED DESCRIPTION:
The study will include 150 patients scheduled to undergo pulmonary vein (PV) ablation because of non-responsive to medical therapy PAF. ECG recordings will be obtained during sinus rhythm before and after PV ablation with a 3 - channel digital recorder for 10 minutes, and digitized with a 16-bit accuracy at a sampling rate of 1000 Hz. The P wave will be analyzed using the Morlet wavelet. Other parameters to be analyzed include 12 lead surface ECG, the burden of main and secondary morphologies and echocardiographic indexes of left atrial mechanical function. Follow-up visits will be held in 3, 6 and 12 months after the ablation procedure.

ELIGIBILITY:
Inclusion Criteria:

* Males and Females
* Age >18 years
* Paroxysmal AF (PAF) scheduled to undergo pulmonary vein (PV) ablation
* Singed written consent form
* Patients who will comply with study procedures

Exclusion Criteria:

* Age <18 years Permanent atrial fibrillation
* Acute myocardial infraction, coronary artery bypass graft surgery or percutaneous transluminal coronary angioplasty within less than 2 months prior to ablation procedure
* Life expectancy less than 12 months, according to investigator's judgment
* Participation to other clinical trial
* Patients who will not be compliant with study procedures

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with paroxysmal atrial fibrillation
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2019-02 (Estimated); Study Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
Number of Paroxysmal Atrial Fibrillation (PAF) relapse(s) | 12 months
  Primary end point is one or more PAF relapse(s) during a period of 12 months after the ablation procedure.

SECONDARY OUTCOMES:
Number of Adverse Events | 12 months
  Adverse Events occurred during study period

CONTACTS AND LOCATIONS:
Overall Officials: Vassilios P Vassilikos, MD, FACC, Study Chair — Aristoteleion University of Thessaloniki, Hippokrateion Hospital
Locations (1):
- Hippokrateion University Hospital, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pappone C, Rosanio S, Oreto G, Tocchi M, Gugliotta F, Vicedomini G, Salvati A, Dicandia C, Mazzone P, Santinelli V, Gulletta S, Chierchia S. Circumferential radiofrequency ablation of pulmonary vein ostia: A new anatomic approach for curing atrial fibrillation. Circulation. 2000 Nov 21;102(21):2619-28. doi: 10.1161/01.cir.102.21.2619. PMID 11085966
- [Background] Liu X, Long D, Dong J, Hu F, Yu R, Tang R, Fang D, Hao P, Lu C, Liu X, He X, Liu X, Ma C. Is circumferential pulmonary vein isolation preferable to stepwise segmental pulmonary vein isolation for patients with paroxysmal atrial fibrillation? Circ J. 2006 Nov;70(11):1392-7. doi: 10.1253/circj.70.1392. PMID 17062959
- [Background] Ouyang F, Antz M, Ernst S, Hachiya H, Mavrakis H, Deger FT, Schaumann A, Chun J, Falk P, Hennig D, Liu X, Bansch D, Kuck KH. Recovered pulmonary vein conduction as a dominant factor for recurrent atrial tachyarrhythmias after complete circular isolation of the pulmonary veins: lessons from double Lasso technique. Circulation. 2005 Jan 18;111(2):127-35. doi: 10.1161/01.CIR.0000151289.73085.36. Epub 2004 Dec 27. PMID 15623542
- [Background] Oral H. Mechanisms of atrial fibrillation: lessons from studies in patients. Prog Cardiovasc Dis. 2005 Jul-Aug;48(1):29-40. doi: 10.1016/j.pcad.2005.06.003. PMID 16194690
- [Background] Pappone C, Santinelli V, Manguso F, Vicedomini G, Gugliotta F, Augello G, Mazzone P, Tortoriello V, Landoni G, Zangrillo A, Lang C, Tomita T, Mesas C, Mastella E, Alfieri O. Pulmonary vein denervation enhances long-term benefit after circumferential ablation for paroxysmal atrial fibrillation. Circulation. 2004 Jan 27;109(3):327-34. doi: 10.1161/01.CIR.0000112641.16340.C7. Epub 2004 Jan 5. PMID 14707026
- [Background] Xia Y, Hertervig E, Kongstad O, Ljungstrom E, Platonov P, Holm M, Olsson B, Yuan S. Deterioration of interatrial conduction in patients with paroxysmal atrial fibrillation: electroanatomic mapping of the right atrium and coronary sinus. Heart Rhythm. 2004 Nov;1(5):548-53. doi: 10.1016/j.hrthm.2004.07.016. PMID 15851217
- [Background] Byrd GD, Prasad SM, Ripplinger CM, Cassilly TR, Schuessler RB, Boineau JP, Damiano RJ Jr. Importance of geometry and refractory period in sustaining atrial fibrillation: testing the critical mass hypothesis. Circulation. 2005 Aug 30;112(9 Suppl):I7-13. doi: 10.1161/CIRCULATIONAHA.104.526210. PMID 16159868
- [Background] Van Beeumen K, Houben R, Tavernier R, Ketels S, Duytschaever M. Changes in P-wave area and P-wave duration after circumferential pulmonary vein isolation. Europace. 2010 Jun;12(6):798-804. doi: 10.1093/europace/eup410. Epub 2010 Jan 3. PMID 20047928
- [Background] Blanche C, Tran N, Rigamonti F, Burri H, Zimmermann M. Value of P-wave signal averaging to predict atrial fibrillation recurrences after pulmonary vein isolation. Europace. 2013 Feb;15(2):198-204. doi: 10.1093/europace/eus251. Epub 2012 Aug 31. PMID 22941968
- [Background] Morlet D, Peyrin F, Desseigne P, Touboul P, Rubel P. Wavelet analysis of high-resolution signal-averaged ECGs in postinfarction patients. J Electrocardiol. 1993 Oct;26(4):311-20. doi: 10.1016/0022-0736(93)90052-f. PMID 8228720
- [Background] Vassilikos V, Dakos G, Chatzizisis YS, Chouvarda I, Karvounis C, Maynard C, Maglaveras N, Paraskevaidis S, Stavropoulos G, Styliadis CI, Mochlas S, Styliadis I. Novel non-invasive P wave analysis for the prediction of paroxysmal atrial fibrillation recurrences in patients without structural heart disease: a prospective pilot study. Int J Cardiol. 2011 Dec 1;153(2):165-72. doi: 10.1016/j.ijcard.2010.08.029. Epub 2010 Sep 15. PMID 20837368
- [Background] Camm AJ, Lip GY, De Caterina R, Savelieva I, Atar D, Hohnloser SH, Hindricks G, Kirchhof P; ESC Committee for Practice Guidelines (CPG). 2012 focused update of the ESC Guidelines for the management of atrial fibrillation: an update of the 2010 ESC Guidelines for the management of atrial fibrillation. Developed with the special contribution of the European Heart Rhythm Association. Eur Heart J. 2012 Nov;33(21):2719-47. doi: 10.1093/eurheartj/ehs253. Epub 2012 Aug 24. No abstract available. PMID 22922413
- [Background] Martinez A, Alcaraz R, Rieta JJ. Application of the phasor transform for automatic delineation of single-lead ECG fiducial points. Physiol Meas. 2010 Nov;31(11):1467-85. doi: 10.1088/0967-3334/31/11/005. Epub 2010 Sep 24. PMID 20871135
- [Background] Packer DL, Kowal RC, Wheelan KR, Irwin JM, Champagne J, Guerra PG, Dubuc M, Reddy V, Nelson L, Holcomb RG, Lehmann JW, Ruskin JN; STOP AF Cryoablation Investigators. Cryoballoon ablation of pulmonary veins for paroxysmal atrial fibrillation: first results of the North American Arctic Front (STOP AF) pivotal trial. J Am Coll Cardiol. 2013 Apr 23;61(16):1713-23. doi: 10.1016/j.jacc.2012.11.064. Epub 2013 Mar 21. PMID 23500312
- [Background] Ketels S, Houben R, Van Beeumen K, Tavernier R, Duytschaever M. Incidence, timing, and characteristics of acute changes in heart rate during ongoing circumferential pulmonary vein isolation. Europace. 2008 Dec;10(12):1406-14. doi: 10.1093/europace/eun287. Epub 2008 Oct 19. PMID 18936041